CLINICAL TRIAL: NCT05748158
Title: Physiology of the Weight Reduced State
Brief Title: A Study to Investigate Why Overweight People Regain Weight After Losing Weight in a Behavioral Weight Loss Program
Acronym: POWERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Tufts University (Other); Columbia University (Other); New York State Psychiatric Institute (Other); Drexel University (Other); University of Pennsylvania (Other); Dartmouth College (Other)
Responsible Party: Principal Investigator, Steven Belle, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY21120046; U24DK128125 (NIH); UH3DK128302 (NIH); UH3DK128298 (NIH)
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Weight change trajectory; Lifestyle intervention
MeSH Terms: conditions — Obesity; Weight Loss; Body-Weight Trajectory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight loss (Other): A 37 week behavioral intervention aimed at decreasing energy intake and increasing physical activity.
  Interventions: Behavioral: Weight loss

INTERVENTIONS:
Behavioral: Weight loss — A behavioral lifestyle program, up to 20 weeks in duration, based on interventions shown to be successful for weight loss such as the Diabetes Prevention Program (DPP), Action for Health in Diabetes (Look AHEAD), and Comprehensive Assessment of the Long-term Effects of Reducing Intake of Energy Study (CALERIE). Weekly sessions, led by experienced interventionists, will provide education and behavioral strategies for weight loss focused an energy-reduced diet and physical activity.
  Participants must meet the following milestones to continue in the study:
  * ≥ 2% weight loss anytime between 28 and 34 days after the start of the intervention
  * ≥ 5% weight loss anytime between 140 and 146 days after the start of the intervention
  * ≥ 7% weight loss by the end of 35 weeks
  After achieving ≥7% weight loss followed by weight stability, participants are observed, without further intervention, for 52 weeks.

SUMMARY:
The goal of this clinical trial is to determine the physiological basis for the differences in weight regain among adults (25-59 years old) with obesity following participation in a behavioral weight loss program. Eligible participants will undergo a baseline evaluation after which they will enter an up to 20 week behavioral weight loss program with the goal of losing at least 7 percent of their baseline weight within 35 weeks. Participants who meet the weight loss goal will be asked to remain weight stable for 2 weeks after which they will undergo a clinical examination. They will then be observed for 1 year during which they will undergo 2 additional clinical examinations, one 4 months after completing the weight loss program, and the other 12 months after completing the weight loss program.

DETAILED DESCRIPTION:
Primary Hypothesis:

Changes, integrated values and patterns in energy intake (EI), energy expenditure (EE), resting energy expenditure (REE) and non-resting energy expenditure (NREE), contribute to the variability in weight change during the 12 months following weight loss.

Assessment time points:

* Baseline (BL): prior to starting the weight loss intervention
* T0: at the end of a period of weight stabilization following at least 7 percent weight loss
* T4: four months (17 weeks) following T0
* T12: twelve months (52 weeks) following T0

Secondary Hypotheses:

Changes, integrated values and patterns in components of EI and EE (listed below) contribute to variability in weight change during the 12 months following weight loss.

EI:

* Psychosocial, food attitude, and food environment assessments
* Diet composition
* Neural activation in food choice/decision-making and cue/taste/reward (functional magnetic resonance imaging [fMRI])
* Measures of food choice, delay discounting, and eating in the absence of hunger
* Gastric emptying, appetite-related peptides, and glucose and lipid excursions in response to a meal

EE:

* Physical activity
* 24-hour urine catecholamine
* Muscle contractile efficiency
* Mitochondrial function in biopsied skeletal muscle
* Sleep quality and patterns

  * Muscle and adipose tissue gene expression
  * Plasma metabolome, proteome, exosomes and exposome
  * Stool microbiome

Specific Aims:

Specific Aim 1: Examine total energy expenditure (TEE) and energy intake (EI) at, and between, baseline, the end of the weight stabilization period following at least 7 percent weight loss, 17 weeks and 52 weeks after the end of the weight stabilization period following at least 7 percent weight loss with respect to variability in weight change between the end of the weight stabilization period following at least 7 percent weight loss and 52 weeks after the end of the weight stabilization period following at least 7 percent weight loss.

Specific Aim 2: Examine resting energy expenditure (REE) and non-resting energy expenditure (NREE) at, and between, baseline, the end of the weight stabilization period following at least 7 percent weight loss, 17 weeks and 52 weeks after the end of the weight stabilization period following at least 7 percent weight loss with respect to variability in weight change between the end of the weight stabilization period following at least 7 percent weight loss and 52 weeks after the end of the weight stabilization period following at least 7 percent weight loss.

Specific Aim 3: Assess endophenotypes of EI (e.g. diet composition, food-choice, decision-making, delay discounting, cue/taste reward, gastric emptying, appetite-related peptides, glucose and lipid excursions in response to a meal, sleep patterns, food and social environments) at and between time points at which they are measured (e.g., baseline, the end of the weight stabilization period following at least 7 percent weight loss, 17 weeks and 52 weeks after the end of the weight stabilization period following at least 7 percent weight loss) and examine their contributions to the variability in weight change between the end of the weight stabilization period following at least 7 percent weight loss and 52 weeks later.

Specific Aim 4: Assess endophenotypes of EE (e.g., actigraphy measures, sleep patterns, muscle contractile efficiency, mitochondrial function, muscle and adipose tissue gene expression, plasma metabolome, microbiome, exposome, and environment) at, and between, time points at which they are measured (e.g., baseline, the end of the weight stabilization period following at least 7 percent weight loss, 17 weeks and 52 weeks after the end of the weight stabilization period following at least 7 percent weight loss) and examine their contributions to the variability in weight change between the end of the weight stabilization period following at least 7 percent weight loss and 52 weeks later.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 25 - <60 years
2. BMI: 30 - <40 kg/m2 at the first screening visit
3. Within 5% of current weight, for the past 6 months at the first screening visit
4. Able to participate in ergometry testing
5. Has a smart phone, tablet or computer with access to the internet

Exclusion Criteria:

1. If 25-29 years old, > 5% deviation from maximum weight (excluding weights while pregnant) since age 25 years
2. If at least 30 years old, > 5% deviation from maximum weight (excluding weights while pregnant) in last 5 years or ≥ 10% deviation from maximum weight (excluding weights while pregnant) since age 30 years
3. History of pulmonary embolus in the past 6 months
4. Cardiovascular disease (e.g. myocardial infarction, stroke, hospitalization for unstable angina, or transient ischemic attack) within the past 6 months
5. Current major depressive disorder or history of major depressive disorder within 2 years
6. Any regular tobacco or nicotine use in the past year
7. Currently engaging in intense physical training or training for a sports event including, but not limited to, a marathon or body building
8. Currently pregnant, or less than one-year post-partum or actively planning to become pregnant within the next two years
9. Presently classified as being in New York Heart Association Class II or greater or dysrhythmia
10. Diabetes (type 1 or 2 - HbA1c ≥ 6.5%, fasting glucose ≥ 126 mg/dL) or currently taking a glucose lowering medication
11. Thyroid disease requiring hormones or medication or TSH < 0.5 or > 5 mIU/L
12. Renal disease requiring dialysis
13. Known HIV infection
14. ALT or AST greater than 5 times the upper limit of normal or active gall bladder disease
15. Significant anemia (Hgb < 10 g/dL) or thrombocytopenia (platelet count < 60,000 /mm3)
16. Leukopenia defined as:

    Males: WBC < 3,100 /mm3 or (WBC 3,100 - < 4,000 /mm3 and at least 1 Duffy antigen (A, B) positive or no result) Females: WBC < 3,400 /mm3 or (WBC 3,400 - < 4,000 /mm3 and at least 1 Duffy antigen (A, B) positive or no result)
17. Active cancer or current chemotherapy treatment, or history of cancer requiring treatment in the past 5 years except for non-melanoma skin cancers or cancers that have clearly been cured
18. Current or past history of anorexia nervosa or bulimia nervosa
19. Current or past diagnosis of binge eating disorder
20. Diagnosis of other severe psychiatric disorder (e.g. schizophrenia, bipolar disorder)
21. Unwillingness to abstain from marijuana/cannabis use for 3 weeks at each of the four assessment time points
22. Known or suspected abuse or misuse of alcohol, prescription drugs, or recreational drugs
23. Antiretroviral therapy (ART), including treatment for HIV, pre-exposure prophylaxis (PrEP) or post-exposure prophylaxis (PEP) within the past 3 months
24. Regularly taking medication or supplement known to affect appetite, energy expenditure, or weight (e.g. appetite suppressants, steroids-including inhaled steroids but not topical, alpha-blockers, beta-blockers, certain psychotropic medications)
25. Currently taking anticoagulant medication
26. Currently enrolled in a supervised weight reduction program
27. Prior or planned bariatric surgery, endoscopic therapy, device-based therapy for obesity, liposuction, cryolipolysis, or abdominoplasty
28. Severely restricted diets: Vegan (no meat, fish, dairy, eggs, or honey), very low carbohydrate (<15% calorie as carbohydrate), very low fat (<15% calories as fat), or strictly gluten free
29. Current celiac or diagnosed gluten intolerance or inflammatory bowel disease requiring specialized diet
30. Night or rotating shift worker
31. Known severe allergy (e.g. anaphylaxis) to nuts or other foods
32. Systolic blood pressure (BP) <90 mmHg and/or diastolic BP <60 mmHg on 2 measurements during the clinical screening visit.
33. Systolic blood pressure (BP) >160 mmHg and/or diastolic BP >100 mmHg on at least 2 measurements during the clinical screening visit or resting heart rate < 45 beats per minute or >100 on 2 measurements during the clinical screening visit.
34. Metal implants, piercings that cannot be removed, or metal-based tattoos or hair treatments
35. Exceeds limitations to fit dual-energy X-ray absorptiometry (DXA) field of view
36. Known allergy to lidocaine or acetaminophen
37. Non-compliance with appointments or tasks (food diaries, etc.) during the screening phase
38. Blood clotting disorder or INR > ULN or PT > ULN or (a)PTT > ULN
39. Tendency to form thick or raised scars
40. Inability to achieve weight stability (defined in section 4.2.1) during the 2 weeks prior to initiation of the baseline Doubly Labeled Water (DLW) assessment
41. At high risk for suicide, as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 205 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Weight change from end of weight stabilization following at least 7 percent weight loss to 52 weeks after weight stabilization following at least 7 percent weight loss | End of weight stabilization following at least 7 percent weight loss vs. 52 weeks after weight stabilization following at least 7 percent weight loss
  Percentage of lost weight that is regained
Weight change from end of weight stabilization following at least 7 percent weight loss to 52 weeks after weight stabilization following at least 7 percent weight loss | End of weight stabilization following at least 7 percent weight loss vs. 52 weeks after weight stabilization following at least 7 percent weight loss
  Weight regained

CONTACTS AND LOCATIONS:
Overall Officials: Steven Belle, PhD, Principal Investigator — University of Pittsburgh; Dympna Gallagher, EdD, Principal Investigator — Columbia University; Susan Roberts, PhD, Principal Investigator — Dartmouth College
Locations (3):
- United States (3):
  - Columbia University Irving Medical Center, New York, New York
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Relevant individual participant data (IPD) will be provided to approved ancillary study investigators. All data will be archived, following the end of the study, at the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)-supported data repository.
Supporting Information: Study Protocol
Time Frame: Following the end of data collection. Time frame is determined by the NIDDK.
Access Criteria: Access to the data for approved ancillary studies will be through the data coordinating center. Access to the data at the NIDDK-repository will be through the NIDDK data repository's process.
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- See also: The Physiology of the Weight Reduced State (POWERS) study website — http://www.powers-study.org/